CLINICAL TRIAL: NCT06345443
Title: The Effect of Oral Nicotinamide Riboside on Systemic Vascular Perfusion in Healthy Adults: A Critical Foundation of Cerebrovascular Health, Cardiovascular Health, and Healthy Aging
Brief Title: NRM on Vascular Perfusion in Healthy Adults
Acronym: NRM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ryan T. Hurt, M.D., Ph.D., Principle Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 23-005288
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Vascular Stiffness
Keywords: cardiovascular; Nicotinamide Riboside; Supplements; NRM

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The pharmacy will be responsible for randomization and dispensing appropriate randomized intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 830 mg Nicotinamide and Placebo (Active Comparator): 830 mg Nicotinamide supplement capsule and 1 identical Placebo capsule twice a day for 12 weeks
  Interventions: Dietary Supplement: Nicotinamide Riboside Malate; Other: Placebo
- 1660 mg Nicotinamide (Active Comparator): 1660 mg Nicotinamide supplement; 2 of the 830 mg capsules twice a day for 12 weeks
  Interventions: Dietary Supplement: Nicotinamide Riboside Malate
- Placebo (Placebo Comparator): 2 identical Placebo capsules twice a day for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside Malate — Active supplement.
  Other Names: NRM
  Arms: 1660 mg Nicotinamide; 830 mg Nicotinamide and Placebo
Other: Placebo — Placebo
  Arms: 830 mg Nicotinamide and Placebo; Placebo

SUMMARY:
The purpose of this study is to better understand the effects of nicotinamide riboside supplement in overall cardiovascular health in healthy adults.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, parallel-dose clinical trial. Participants will be randomly assigned to one of three groups. Study measurements will be completed at three timepoints and intervention taken daily throughout the subject's 12 weeks of participation.

ELIGIBILITY:
Inclusion Criteria:

* >= 40 and <=60
* Provides consent to participate in the study
* Not pregnant at time of consent
* Understands and agrees to follow all study procedures and limitations
* Have no contraindicating comorbid health condition as determined by the clinical investigators

Exclusion Criteria:

* Pregnant, nursing, or trying to conceive
* BMI Restrictions: <30
* Allergy or sensitivity to study agent ingredients
* Hypertension treated with medication
* Use of natural health products containing nicotinamide riboside, quercetin, trans-resveratrol, or betaine anhydrous within 7 days prior to randomization and during the course of the study.
* Surgery planned during the course of the trial
* History or past diagnosis of chronic diseases, unstable medical conditions, blood/bleeding disorders or stroke
* History or current diagnosis of cancer (except for successfully treated basal cell carcinoma diagnosed less than 5 years prior to screening or cancer in full remission more than 5 years after diagnosis.
* Abnormal blood chemistries for renal or liver function (defined as 1 standard deviation outside of the normal range), alcohol dependence, uncontrolled thyroid disease, severe obesity (body mass index >40 kg m-2), or weight stable for at least 3 months prior to enrolling in the study (defined as >2 kg change in body mass).
* An unstable medical or mental health condition as determined by the physician investigator.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Reduced Endothelial Stiffness | Baseline to End of study at 12 weeks
  Endothelial Peripheral Arterial Tonometry testing will be used to assess endothelial stiffness changes over study

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hurt, MD, PhD, Principal Investigator — Mayo Clinic; Brent Bauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No